CLINICAL TRIAL: NCT02067325
Title: Effects of Thai Massage on EMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Vitsarut Buttagat, Dr. Vitsarut Buttagat, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55218152-2
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Medicine, Thai Traditional

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thai massage (Experimental): The participants will receive thirty minutes session of Thai massage onto the trapezius muscle for 1 sessions
  Interventions: Other: Thai massage
- Sham Microwave diathermy (Sham Comparator): The participants will receive thirty minutes session of Sham Microwave diathermy onto the trapezius muscle for 1 sessions
  Interventions: Other: Thai massage

INTERVENTIONS:
Other: Thai massage

SUMMARY:
The purpose of this study is to determine the effect of Thai massage on electromyogram in patients with chronic upper back pain associated with myofascial trigger points.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age between 18 - 50 years old
* The participants have experienced spontaneous upper pain for longer than 12 weeks (chronic) and that at least one trigger point will be present in the s trapezius muscles. Trigger points will be diagnosed as the presence of focal tenderness in a taut band and with pain recognition.
* The participants will be able to follow instructions.
* Good communication and cooperation.

Exclusion Criteria:

* A history of the following diseases or disorders:
* Cervical radiculopathy
* Contraindications of traditional Thai massage
* Contagious skin disease
* Injury or inflammation of muscle
* Bone fracture and/or joint dislocation
* Open wound
* Uncontrolled hypertension
* Drug and/or alcohol intoxication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Muscle activity as a Measure of Electromyogram | 1 day

SECONDARY OUTCOMES:
Pain scores on Visual Analog Scale | 1 day
Muscle tension on Visual Analog Scale | 1 days

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Science, Mae Fah Luang University, Mueang, Changwat Chiang Rai, Thailand

REFERENCES:
- [Derived] Buttagat V, Narktro T, Onsrira K, Pobsamai C. Short-term effects of traditional Thai massage on electromyogram, muscle tension and pain among patients with upper back pain associated with myofascial trigger points. Complement Ther Med. 2016 Oct;28:8-12. doi: 10.1016/j.ctim.2016.07.004. Epub 2016 Jul 19. PMID 27670864